CLINICAL TRIAL: NCT00232830
Title: Trial to Assess the Use of the Cypher TM Stent in Acute Myocardial Infarction Treated With Balloon Angioplasty
Brief Title: The Study to Assess AMI Treated With Balloon Angioplasty.
Acronym: TYPHOON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans-Peter Stoll, Cordis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC03-03
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cypher Sirolimus-eluting Coronary Stent
  Interventions: Device: drug-eluting stent
- 2 (Active Comparator): Bare-metal stent
  Interventions: Device: bare-metal stent

INTERVENTIONS:
Device: drug-eluting stent — Cypher Sirolimus-eluting Coronary Stent
  Arms: 1
Device: bare-metal stent — any bare-metal stent brand
  Arms: 2

SUMMARY:
The main objective of this study is to assess the effectiveness and safety of the CYPHER™ (CYPHER SELECT™) (Sirolimus-eluting) stent in reducing the occurrence of a composite endpoint of target vessel failure (TVF) in subjects treated for acute myocardial infarction as compared to a bare metal stent.

DETAILED DESCRIPTION:
This is an international, multicenter (up to 52 sites), randomized, single-blind study in patients with an acute myocardial infarction treated with the CYPHER™ (Sirolimus-eluting) stent as compared to the bare stents.

Patients with de novo native coronary artery lesions will be treated with the CYPHER™ (Sirolimus-eluting) stent or a bare stent. Subjects will be followed at 30 days, 6 months and at 1, 3, 4 and 5 years post-procedure. 200 subjects will have an angiographic follow-up at 8 months.

ELIGIBILITY:
Inclusion Criteria:

1. Have prolonged, continuous (lasting at least 20 minutes) chest pain despite administration of nitrates and onset within 12 hours of randomization, and one of the following:

   1. ST segment elevation >=1mm in standard leads and >=2mm in 2 or more contiguous precordial leads with reciprocal ST depression
   2. New or presumably new left bundle branch block (LBBB)
2. The culprit lesion must be identified on a de novo native coronary artery and an emergency angioplasty must be possible. The culprit site must be visualized before the stent implantation;

Exclusion Criteria:

1. Killip class > 2 upon arrival to the cath-lab;
2. Significant (>50%) stenosis proximal or distal to the target lesion that might require revascularization or impede inflow or runoff;
3. Evidence of massive thrombus in the infarct related artery distally to the culprit lesion;
4. Documented left ventricular ejection fraction <=30%;
5. Target lesion is located in an arterial or venous by-pass graft;
6. ECG documented evidence of prior myocardial infarction;
7. Patient who received thrombolytic therapy for the current AMI before enrollment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 715 (Actual)
Dates: Start 2003-10; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Composite of target vessel failure (TVF) defined as target vessel revascularization, recurrent myocardial infarction, or cardiac death that could not be clearly attributed to a vessel other than the target vesselpost-procedure. | 1 and 6 months and at 1, 3, 4, and 5 years post-procedure.

SECONDARY OUTCOMES:
cardiac death | 1, 3, 4 and 5 years post-procedure
recurrence of myocardial infarction | 1, 3, 4 and 5 years post-procedure
revascularization of the target vessel (TVR) | 1, 3, 4 and 5 years post-procedure
recurrence of ischemia | 1, 3, 4 and 5 years post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Christian Spaulding, MD, Principal Investigator — HOPITAL COCHIN, René Descartes University; Christoph Bode, MD, Principal Investigator — University of Freiburg, Albert-Ludwigs-Universitätskliniken
Locations (2):
- HOPITAL COCHIN, René Descartes University, Paris, France
- University of Freiburg, Albert-Ludwigs-Universitätskliniken, Freiburg im Breisgau, Germany

REFERENCES:
- [Result] Spaulding C, Henry P, Teiger E, Beatt K, Bramucci E, Carrie D, Slama MS, Merkely B, Erglis A, Margheri M, Varenne O, Cebrian A, Stoll HP, Snead DB, Bode C; TYPHOON Investigators. Sirolimus-eluting versus uncoated stents in acute myocardial infarction. N Engl J Med. 2006 Sep 14;355(11):1093-104. doi: 10.1056/NEJMoa062006. PMID 16971716
- [Result] Rozenman Y, Witzling V, Tamari I, Turkisher V, Kriviski M, Bode C, Henry P, Teiger E, Cebrian A, Stoll HP, Spaulding C. Impact of stent length on restenosis in patients with acute myocardial infarction treated with primary percutaneous coronary intervention: analysis based on data from the Trial to Assess the Use of the Cypher Stent in Acute Myocardial Infarction Treated with Balloon Angioplasty (TYPHOON). EuroIntervention. 2009 Jun;5(2):219-23. doi: 10.4244/eijv5i2a34. PMID 19527979
- [Derived] Spaulding C, Teiger E, Commeau P, Varenne O, Bramucci E, Slama M, Beatt K, Tirouvanziam A, Polonski L, Stella PR, Clugston R, Fajadet J, de Boisgelin X, Bode C, Carrie D, Erglis A, Merkely B, Hosten S, Cebrian A, Wang P, Stoll HP, Henry P. Four-year follow-up of TYPHOON (trial to assess the use of the CYPHer sirolimus-eluting coronary stent in acute myocardial infarction treated with BallOON angioplasty). JACC Cardiovasc Interv. 2011 Jan;4(1):14-23. doi: 10.1016/j.jcin.2010.10.007. PMID 21251624